CLINICAL TRIAL: NCT06300879
Title: A Prospective Study on the Perioperative Safety and Short-Term Quality of Life in Totally Laparoscopic Proximal Gastrectomy With Esophagogastrostomy by Fissure Technique
Brief Title: A Prospective Study on Esophagogastrostomy by an Innovative Surgical Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Hao Hankun, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1058
Record Dates: First submitted 2024-02-18; First posted 2024-03-08 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Gastric Cancer; Adenocarcinoma of Esophagogastric Junction
Keywords: proximal gastrectomy; totally laparoscopic gastrectomy; fissure technique
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients included in this group will receive totally laparoscopic proximal gastrectomy with esophagogastrostomy by fissure technique，which is an innovative surgery that investigators first began to apply in patients with proximal gastric cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): Performing totally laparoscopic proximal gastrectomy with esophagogastrostomy by fissure technique
  Interventions: Procedure: Performing totally laparoscopic proximal gastrectomy with esophagogastrostomy by fissure technique

INTERVENTIONS:
Procedure: Performing totally laparoscopic proximal gastrectomy with esophagogastrostomy by fissure technique — Surgical Operation:
  1. Gastric Resection Range:Proximal gastrectomy, preserving 2/3 of the distal stomach.
  2. Lymph Node Dissection Range:D1+ to D2 lymph node dissection.
  3. Anastomosis Method: esophagogastrostomy by fissure technique.
  4. Anastomosis Risk Management Plan:For a rupture with a maximum diameter less than or equal to 5mm, repair with 4-0/3-0 absorbable sutures and proceed with the anastomosis.For a rupture with a maximum diameter greater than 5mm or failed anastomosis, resect that part of the remaining stomach, change to proximal gastrectomy, and perform double-channel anastomosis.
  5. Surgical Approach:Totally laparoscopic proximal gastrectomy.

SUMMARY:
This is a single-center, open-label, Phase Ib/II study aiming to assess the perioperative safety and postoperative outcomes of a novel surgical technique in treating primary adenocarcinoma located in the upper 1/3 of the stomach or gastroesophageal junction (Siewert II or III).

The study will enroll 30 patients who will undergo totally laparoscopic proximal gastrectomy with esophagogastrostomy by fissure technique. Clinical data will be collected to evaluate perioperative safety. Patients will be followed for at least 3 months, during which endoscopy will be performed to analyze occurrences and reasons for anastomotic-related complications. Additionally, the quality of life after surgery will be evaluated by QLQ-C30 and QLQ-STO22.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old;
2. Pathologically confirmed as adenocarcinoma;
3. Primary tumor located in the upper 1/3 of the stomach or the gastroesophageal junction (Siewert II or III);
4. If it is adenocarcinoma of the upper 1/3 of the stomach, cT1N0M0 should be met.
5. For gastroesophageal junction adenocarcinoma, cT1-2N0M0 should be met, and clinical judgment should indicate no distant lymph node metastasis around the stomach.
6. Bilateral resection margins should be greater than 2 cm, and more than half of the residual stomach should be preserved.
7. No history of upper abdominal surgery (excluding laparoscopic cholecystectomy).
8. No preoperative comprehensive treatments such as chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc.
9. Preoperative ECOG (Eastern Cooperative Oncology Group) score of 0/1.
10. Preoperative ASA (American Society of Anesthesiologists) score I-III.
11. Good function of important organs.
12. Signed informed consent.

Exclusion Criteria:

1. Preoperative assessment indicating cT4b or Bulky lymph nodes enlargement or distant lymph nodes metastasis;
2. Pregnant or lactating women;
3. Patients with severe mental illness;
4. Preoperative temperature ≥38°C or infectious diseases requiring systemic treatment;
5. Severe respiratory diseases, with FEV1 < 50% of predicted value;
6. History of other malignant tumors in the past 5 years;
7. Severe liver or kidney dysfunction;
8. Unstable angina or myocardial infarction within the last 6 months;
9. History of stroke or cerebral hemorrhage within the last 6 months (excluding old infarcts);
10. Systemic use of glucocorticoids within the last 1 month;
11. Emergency surgery required due to complications of gastric cancer (bleeding, perforation, obstruction);
12. Patient has participated in or is currently participating in other clinical trials (within the last 6 months).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Assess intraoperative Perioperative Safety by Duration of surgery. | intraoperative
  Time spent on the whole operation（minutes）
Assess intraoperative Perioperative Safety by Duration of anastomosis. | intraoperative
  Time spent on the anastomosis in minutes
Assess intraoperative Perioperative Safety by blood loss . | intraoperative
  Intraoperative blood loss in milliliters
Postoperative recovery course | 30 days after the surgery
  Time to remove the drain tube,flatus, to liquid diet, and soft diet are used to assess the postoperative recovery course, which is a composite outcome measure.
Postoperative TNM staging by Pathological findings . | 30 days after the surgery
  AJCC（American Joint Committee on Cancer）-8th TNM staging system will be used to obtain pathology of tumor .

SECONDARY OUTCOMES:
The incidence of postoperative reflux esophagitis | 3 months after surgery
  Patients will be monitored for the incidence of postoperative reflux esophagitis after surgery by weight changes, blood biochemistry and endoscopic examination
The incidence of postoperative anastomotic stenosis | 3 months after surgery
  Patients will be monitored for the incidence of postoperative reflux esophagitis after surgery by weight changes, blood biochemistry and endoscopic examination
Quality of Life at 3 Months Postoperatively will be assessed by EORTC QLQ-C30 | 3 months after surgery
  QLQ-C30 is a comprehensive assessment of the overall quality of life dimensions before and after surgery for patients. Higher scores represent poorer quality of life for patients after surgery.
Quality of Life at 3 Months Postoperatively will be assessed by EORTC QLQ-STO22 scale | 3 months after surgery
  QLQ-STO22 is a specific assessment for postoperative situations related to anastomosis, such as swallowing and eating.Higher scores represent poorer quality of life for patients after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No